CLINICAL TRIAL: NCT06547710
Title: Primary Tumor Resection for M1a Stage Lung Cancer With Occult Pleural Dissemination Discovered During Surgery: a Prospective, Single-arm, Multi-center, Phase Ⅱ Trial
Brief Title: Primary Tumor Resection for M1a Stage Lung Cancer
Acronym: ECTOP-1023
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director of Thoracic Surgery Department, Fudan University
Other Study IDs: ECTOP-1023
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer Metastatic; Surgical Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1023. This study aims to explore the safety and efficacy of primary lesion resection in the treatment of M1a stage lung cancer with pleural dissemination found during surgery, and to more accurately evaluate whether primary lesion resection can improve the OS and quality of life of the corresponding patients.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research, willing to follow and able to complete all trial procedures;
2. Aged 18-80 years (including critical values) when signing the informed consent form;
3. ECOG score 0 or 1;
4. No previous lung cancer surgery;
5. Intraoperative or postoperative pathological confirmation of M1a stage lung cancer;
6. Occult pleural metastasis found during surgery;
7. Preoperative lymph node staging is cN0;
8. First-time treatment and no radiotherapy or chemotherapy.

Exclusion Criteria:

1. The lesion cannot be completely removed surgically;
2. Cytological or histological pathology confirms other lung malignancies other than lung cancer;
3. Patients who have undergone lung cancer surgery before;
4. Patients who have received radiotherapy or chemotherapy and are not treatment-naive patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-75
Study Population: This clinical trial is a single-arm, multicenter, prospective, confirmatory phase II clinical study, which mainly evaluates the efficacy and safety of primary lesion resection for patients with M1a stage lung cancer who have occult pleural dissemination during surgery (Figure 1). Since it is unethical not to perform primary lesion resection during surgery for such patients, this study is a single-arm one. Primary lesion resection should be a resection that can completely remove the primary lesion, including lobectomy and sublobar resection.
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Median overall survival | About 10months.
  Median overall survival for M1a patients underging surgery.

SECONDARY OUTCOMES:
2-year overall survival | 2 years
  2-year overall survival
5-year overall survival | 5 years
  5-year overall survival
FEV1 and FVC | 0.5 year
  Preoperative lung function test

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China